CLINICAL TRIAL: NCT01422551
Title: Facilitating Positive Adaptation to Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael H. Antoni, Principle Investigator, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 19930536; R01CA064710 (NIH)
Record Dates: First submitted 2011-08-21; First posted 2011-08-24 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: stress management intervention; breast cancer; quality of life; psychosocial adaptation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Stress Management (Experimental): 10 weekly 2-hour sessions of group-based cognitive behavioral stress management
  Interventions: Behavioral: Cognitive Behavioral Stress Management
- Psycho-educational Control (Active Comparator): a single day group-based psycho-educational seminar
  Interventions: Behavioral: a psycho-educational control

INTERVENTIONS:
Behavioral: Cognitive Behavioral Stress Management — 10 weekly 2-hour sessions of group-based cognitive behavioral stress management
  Arms: Cognitive Behavioral Stress Management
Behavioral: a psycho-educational control — a single-day psycho-educational seminar
  Arms: Psycho-educational Control

SUMMARY:
The purpose of this study is to test the effects of a 10-wk cognitive behavioral stress management (CBSM) intervention vs. a single-day psycho-educational seminar on psychosocial adaptation and physiological adaptation in women being treated for stage I-III breast cancer.

DETAILED DESCRIPTION:
The study tests the effects of a 10-wk group-based cognitive behavioral stress management (CBSM) intervention (relaxation, stress awareness, cognitive restructuring, coping skills training, interpersonal skills training) versus a single-day psycho-educational seminar (general information about stress and coping) in women who have recently had surgery for breast cancer but have not yet started adjuvant therapy. The study evaluates the effects of CBSM on psychosocial adaptation (includes measures of negative adaptation [distress and social disruption] and positive adaptation [benefit finding and positive affect]) at 6-month and 12-month follow-up. The study also evaluates the effects of CBSM on physiological adaptation (includes levels of PM serum cortisol and T-helper-type 1 (Th1) cytokine [interleukin-2, IL-2, and interferon-gamma, IFN-g, production after anti-CD3 stimulation of peripheral blood mononuclear cells (PBMC).

ELIGIBILITY:
Inclusion Criteria:

-women diagnosed with breast cancer at stage III or below who had recently undergone lumpectomy or mastectomy

Exclusion Criteria:

* prior cancer,
* prior psychiatric treatment for a serious disorder (e.g., psychosis, suicidality),
* lack of fluency in English and had begun adjuvant therapy at time of first assessment

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 1999-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
change from baseline to 12 month follow-up in psychosocial adaptation (less negative affect and social disruption; more benefit finding and positive affect) | baseline and 6 and 12 month follow-up
  changes in a composite composed of negative affect measures plus a measure of social disruption plus a measure of benefit finding plus a measure of positive affect

SECONDARY OUTCOMES:
change from baseline to 12 months in physiological adaptation (decreased serum cortisol and increased Th1 cytokine production) | baseline and 6 and 12 months follow-up
  decreased PM levels of serum cortisol and increased Th1 (interleukin-2, interferon-gamma) cytokine production following anti-CD3 stimulation of peripheral blood mononuclear cells (PBMCs)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Antoni, Ph.D., Principal Investigator — University of Miami
Locations (1):
- Department of Psychology University of Miami, Coral Gables, Florida, United States

REFERENCES:
- [Result] Antoni MH, Wimberly SR, Lechner SC, Kazi A, Sifre T, Urcuyo KR, Phillips K, Smith RG, Petronis VM, Guellati S, Wells KA, Blomberg B, Carver CS. Reduction of cancer-specific thought intrusions and anxiety symptoms with a stress management intervention among women undergoing treatment for breast cancer. Am J Psychiatry. 2006 Oct;163(10):1791-7. doi: 10.1176/ajp.2006.163.10.1791. PMID 17012691
- [Result] Antoni MH, Lechner SC, Kazi A, Wimberly SR, Sifre T, Urcuyo KR, Phillips K, Gluck S, Carver CS. How stress management improves quality of life after treatment for breast cancer. J Consult Clin Psychol. 2006 Dec;74(6):1143-52. doi: 10.1037/0022-006X.74.6.1152. PMID 17154743
- [Result] Antoni MH, Lechner S, Diaz A, Vargas S, Holley H, Phillips K, McGregor B, Carver CS, Blomberg B. Cognitive behavioral stress management effects on psychosocial and physiological adaptation in women undergoing treatment for breast cancer. Brain Behav Immun. 2009 Jul;23(5):580-91. doi: 10.1016/j.bbi.2008.09.005. Epub 2008 Sep 20. PMID 18835434
- [Result] Phillips KM, Antoni MH, Lechner SC, Blomberg BB, Llabre MM, Avisar E, Gluck S, DerHagopian R, Carver CS. Stress management intervention reduces serum cortisol and increases relaxation during treatment for nonmetastatic breast cancer. Psychosom Med. 2008 Nov;70(9):1044-9. doi: 10.1097/PSY.0b013e318186fb27. Epub 2008 Oct 8. PMID 18842742
- [Result] Blomberg BB, Alvarez JP, Diaz A, Romero MG, Lechner SC, Carver CS, Holley H, Antoni MH. Psychosocial adaptation and cellular immunity in breast cancer patients in the weeks after surgery: An exploratory study. J Psychosom Res. 2009 Nov;67(5):369-76. doi: 10.1016/j.jpsychores.2009.05.016. Epub 2009 Sep 24. PMID 19837199
- [Derived] Jutagir DR, Blomberg BB, Carver CS, Lechner SC, Timpano KR, Bouchard LC, Gudenkauf LM, Jacobs JM, Diaz A, Lutgendorf SK, Cole SW, Heller AS, Antoni MH. Social well-being is associated with less pro-inflammatory and pro-metastatic leukocyte gene expression in women after surgery for breast cancer. Breast Cancer Res Treat. 2017 Aug;165(1):169-180. doi: 10.1007/s10549-017-4316-3. Epub 2017 May 30. PMID 28560656
- [Derived] Antoni MH, Bouchard LC, Jacobs JM, Lechner SC, Jutagir DR, Gudenkauf LM, Carver CS, Lutgendorf S, Cole SW, Lippman M, Blomberg BB. Stress management, leukocyte transcriptional changes and breast cancer recurrence in a randomized trial: An exploratory analysis. Psychoneuroendocrinology. 2016 Dec;74:269-277. doi: 10.1016/j.psyneuen.2016.09.012. Epub 2016 Sep 24. PMID 27689900
- [Derived] Bouchard LC, Antoni MH, Blomberg BB, Stagl JM, Gudenkauf LM, Jutagir DR, Diaz A, Lechner S, Gluck S, Derhagopian RP, Carver CS. Postsurgical Depressive Symptoms and Proinflammatory Cytokine Elevations in Women Undergoing Primary Treatment for Breast Cancer. Psychosom Med. 2016 Jan;78(1):26-37. doi: 10.1097/PSY.0000000000000261. PMID 26569533
- [Derived] Stagl JM, Bouchard LC, Lechner SC, Blomberg BB, Gudenkauf LM, Jutagir DR, Gluck S, Derhagopian RP, Carver CS, Antoni MH. Long-term psychological benefits of cognitive-behavioral stress management for women with breast cancer: 11-year follow-up of a randomized controlled trial. Cancer. 2015 Jun 1;121(11):1873-81. doi: 10.1002/cncr.29076. Epub 2015 Mar 23. PMID 25809235
- [Derived] Vargas S, Antoni MH, Carver CS, Lechner SC, Wohlgemuth W, Llabre M, Blomberg BB, Gluck S, DerHagopian RP. Sleep quality and fatigue after a stress management intervention for women with early-stage breast cancer in southern Florida. Int J Behav Med. 2014 Dec;21(6):971-81. doi: 10.1007/s12529-013-9374-2. PMID 24318654
- [Derived] Antoni MH, Lutgendorf SK, Blomberg B, Carver CS, Lechner S, Diaz A, Stagl J, Arevalo JM, Cole SW. Cognitive-behavioral stress management reverses anxiety-related leukocyte transcriptional dynamics. Biol Psychiatry. 2012 Feb 15;71(4):366-72. doi: 10.1016/j.biopsych.2011.10.007. Epub 2011 Nov 16. PMID 22088795